CLINICAL TRIAL: NCT05207241
Title: The Guidance on the Gravitationally Assisted Lactation Influences the Occurrence of Lactational Mastitis: a Clinical Cohort Study
Brief Title: The Effect of Gravity on the Occurrence of Lactational Mastitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Jianyi Li, Principal Investigator, Shengjing Hospital
Other Study IDs: Shengjing-LJY05
Record Dates: First submitted 2021-12-21; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Lactation Mastitis
Keywords: Lactation breastfeeding position; mastitis; gravity; breastfeeding position
MeSH Terms: conditions — Mastitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Control group: Under the professional guidance of doctors, participating women (1) breastfeed individually without using a breast pump; (2) massage their breasts 4 times a day for 15 minutes each time; (3) breastfeeding time is scientifically matched with infant's schedule; (4) alternative breastfeed, ensuring emptying one breast within 24 hours. Doctors follow up once a month via WeChat. Participants complete the questionnaires. A breast ultrasound will be performed every three months. The infant weight will be measured and recorded 6 months after breastfeeding
  Interventions: Other: provides guidance on gravitationally assisted breastfeeding

INTERVENTIONS:
Other: provides guidance on gravitationally assisted breastfeeding — Prior to the first breastfeeding after delivery, the guidance of gravitationally assisted breastfeeding will be provided. The primary breastfeeding position is advised to be the sitting position, supplemented by the lateral position with a time ratio of 4:1. The following guidance will also be given: (1) participating women breastfeed individually without using a breast pump; (2) massage their breasts 4 times a day for 15 minutes each time; (3) breastfeeding time is scientifically matched with infant's schedule; (4) alternative breastfeed, ensuring emptying one breast within 24 hours. Doctors follow up once a month via WeChat. Participants complete the questionnaires. A breast ultrasound will be performed every three months. The infant weight will be measured and recorded 6 months after breastfeeding.

SUMMARY:
Lactation is the instinct of almost all mammals, including human beings. With the development of human society, the function of lactation has gradually deviated from nature instinct. Breastfeeding related industries, such as milk bottles, formula and breast pumps, have formed a vast consumer market, leading to a transition from breastfeeding mothers' individual instinct to the social division of labor. Previous studies found that the incidence of lactational mastitis remains largely unchanged post World War II with some reporting an increase, suggesting the hazards of lactational mastitis still exist under the background of social division of labor. Breast milk contains ingredients that improve the immunity of newborns. By affecting mothers' breastfeeding, lactational mastitis pose a hazard for newborns, increasing the chances of developing respiratory and gastrointestinal diseases. For breastfeeding mothers, severe mastitis may develop into breast abscess due to improper treatment in the early stage. In addition to antibiotic treatment, incision, drainage and even surgery may be required. These potentially increase the risk of developing postpartum depression, type II diabetes, breast cancer and ovarian cancer. Compared with other mammals, humans and cows have a higher incidence of lactational mastitis, indicating that human intervention in breastfeeding may be the cause of the high incidence. On the other hand, as a result of walking upright, humans' hands are liberated, forming complex and diverse breastfeeding position. According to the Sakra World Hospital, these positions are classified into eight types: cradle, cross cradle, supine, football, Australian hold, inverted lateral, lateral cradle, and lateral. The pilot study demonstrated that different breastfeeding positions are closed related to the occurrence of lactational mastitis, and to the location of mastitis. Assuming that the baby's sucking factors remain the same, there must be differences in the milk drainage in different breastfeeding positions under the influence of gravity. Researchist speculate that breastfeeding women who opt to a position that cause an anti-gravitational expulsion of milk are more likely to develop lactational mastitis. Therefore, this study aims to investigate how the scientific guidance on the gravitationally assisted breastfeeding positions will reduce the occurrence of mastitis.

DETAILED DESCRIPTION:
Time of recruitment: 1 December 2021 - 30 April 2022. Two thousand women who meet the following criteria are to be recruited:(1) primparious women; (2) full-term delivery;(3) age ≤35 (4) breastfeeding within 7 days after delivery; (5) with autonomous behavior ability; (6) provide voluntary informed consent; (7) ability to breastfeed individually(8) prenatal breast ultrasound shows no breast lesions.. Exclusive criteria: (1) abnormal breast or nipple development (Poland syndrome or degree II and above inverted nipple); (2) history of breast surgery; (3) history of chest radiotherapy; (4) history of malignant tumors; (5) History of mastitis; (6) severe cardiovascular and cerebrovascular diseases, chronic diseases (Ecog score >3, long-term medication affects breastfeeding); (7) skin diseases or connective tissue diseases; (8) Hepatitis, syphilis, gonorrhea, AIDS and other infectious diseases. Criteria of elimination after recruitment: (1) failure to follow the breastfeeding instruction; (2) painless breast mass.

Participants are to be randomly divided into the interventional group which provides guidance on gravitationally assisted breastfeeding, and into the control group which provides general breastfeeding guidance. Through the social media network WeChat, each participant receives breastfeeding guidance before their first breastfeeding, and once a month until 6 months after childbirth. Additionally, at 3 and 6 postpartum, the breasts will be examined by a breast surgeon at Shenyang Women and Infants Hospital. Infant's height and weight will be measured and recorded at 6 months. The incidence of breastfeeding mastitis and the rate of baby weight gain are compared between the groups. This clinical cohort study aims to investigate effects of scientific guidance on the gravitationally assisted breastfeeding positions on the occurrence of breast mastitis.

ELIGIBILITY:
Inclusion Criteria:

* primparious women;
* full-term delivery;
* age ≤35;
* breastfeeding within 7 days after delivery;
* with autonomous behavior ability;
* provide voluntary informed consent; • ability to breastfeed individually;
* prenatal breast ultrasound shows no breast lesions.

Exclusion Criteria:

* abnormal breast or nipple development (Poland syndrome or degree II and above inverted nipple);
* istory of breast surgery;
* history of chest radiotherapy;
* history of malignant tumors;
* history of mastitis;
* severe cardiovascular and cerebrovascular diseases, chronic diseases (Ecog score >3, long-term medication affects breastfeeding);
* skin diseases or connective tissue diseases;
* Hepatitis, syphilis, gonorrhea, AIDS and other infectious diseases.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: * primparious women;
  * full-term delivery;
  * age ≤35;
  * breastfeeding within 7 days after delivery;
  * with autonomous behavior ability;
  * provide voluntary informed consent;
  * ability to breastfeed individually;
  * prenatal breast ultrasound shows no breast lesions.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of lactational mastitis during breastfeeding | Six months
  The incidence of lactational mastitis is defined as the proportion of breastfeeding mastitis that occurs during the period between the first breastfeeding and 6 months post-partum.

SECONDARY OUTCOMES:
Breast swelling and pain | Six months
  Mastitis is caused by the failure of milk to discharge in time, resulting in milk accumulation.Milk accumulation is a prodrome of lactational mastitis.

CONTACTS AND LOCATIONS:
Overall Officials: Jianyi Li, Master, Principal Investigator — Cancer Hospital of China Medical University, Liaoning Cancer Hospital
Locations (1):
- Cancer Hospital of China Medical University, Liaoning Cancer Hospital and Institute, Shenyang, Liaoning, China